CLINICAL TRIAL: NCT02267226
Title: Prospective, Open-label, Uncontrolled, Phase III Study to Assess the Efficacy and Safety of Octafibrin for On-demand Treatment of Acute Bleeding and to Prevent Bleeding During and After Surgery in Subjects With Congenital Fibrinogen Deficiency
Brief Title: Efficacy and Safety Study of Octafibrin for On-demand Treatment of Acute Bleeding and to Prevent Bleeding During and After Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Octapharma (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FORMA-02
Record Dates: First submitted 2014-08-07; First posted 2014-10-17 (Estimated); Results first posted 2019-02-20 (Actual); Last update posted 2021-01-15 (Actual); Status verified 2020-12

CONDITIONS: Congenital Fibrinogen Deficiency

ARMS (1):
- Octafibrin (Experimental)
  Interventions: Drug: Octafibrin

INTERVENTIONS:
Drug: Octafibrin

SUMMARY:
The purpose of the study is to assess the efficacy and safety of Octafibrin for on-demand treatment of acute bleeding in subjects with congenital fibrinogen deficiency.

ELIGIBILITY:
Inclusion Criteria:

* Aged ≥12 years (only 18 and above in Russia)
* Documented diagnosis of congenital fibrinogen deficiency, expected to require on-demand treatment for bleeding or surgical prophylaxis:
* Fibrinogen deficiency manifested as afibrinogenaemia or severe hypofibrinogenaemia.
* Historical plasma fibrinogen activity of <50 mg/dL or levels below the limit of detection of the local assay method.
* Expected to have an acute bleeding episode (spontaneous or after trauma) or planning to undergo elective surgery.
* Informed consent signed by the subject or legal guardian.

Exclusion Criteria:

* Life expectancy <6 months.
* Bleeding disorder other than congenital fibrinogen deficiency, including dysfibrinogenaemia.
* Prophylactic treatment with a fibrinogen concentrate.

Treatment with:

* Any fibrinogen concentrate or other fibrinogen-containing blood product within 2 weeks prior to start of treatment for the bleeding episode or surgery.
* Any coagulation-active drug (i.e., non-steroidal anti-inflammatory drugs, warfarin, coumarin derivatives, platelet aggregation inhibitors) within 1 week prior to start of treatment for the bleeding episode or surgery, or as a planned or expected medication during the time period from Day 1 until 24 hours (i.e., 1 day) after the last Octafibrin infusion.

Presence or history of:

* Hypersensitivity to study medication.
* Deep vein thrombosis or pulmonary embolism within 1 year prior to start of treatment for the bleeding episode or surgery.
* Arterial thrombosis within 1 year prior to start of treatment for the bleeding episode or surgery
* Hypersensitivity to human plasma proteins.
* Oesophageal varicose bleeding.
* End-stage liver disease (i.e., Child-Pugh score B or C).

Pregnant women within the first 20 weeks of gestation.

Currently breast-feeding.

Known positive HIV infection with a viral load >200 particles/μL or >400,000 copies/mL.

Polytrauma 1 year prior to start of treatment for the bleeding episode or surgery.

Diagnosis or suspicion of a neutralizing anti-fibrinogen inhibitor currently or any time in the past.

Acute or chronic medical condition which may, in the opinion of investigator, affect the conduct of the study, including

* Subjects receiving immune-modulating drugs (other than anti-retroviral chemotherapy) such as alpha-interferon, prednisone (equivalent to >10 mg/day), or similar drugs at study start.
* Subjects having evidence or a history (within the previous 12 months) of abuse of any licit or illicit drug substance.

Participation in another interventional clinical study currently or during the past 4 weeks.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2014-09; Primary Completion 2018-02-14 (Actual); Study Completion 2018-02-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Cristina Solomon, MD, Study Director — Octapharma
Locations (12):
- Miami Children's Hospital, Miami, Florida, United States
- Dept of Clinical Hematology for Hemorrhagic Diatheses and Anaemia, SHAT "Joan Pavel", Sofia, Bulgaria
- India (3):
  - St. John's Medical College Hospital, Bangalore
  - Sahyadri Specialty Hospital, Pune
  - Dept of Hematology, Christian Medical College, Vellore
- Iran (2):
  - Seyed Al Shohada Hospital, Isfahan
  - Dastgheib Hospital, Shīrāz
- Hotel-Dieu de France, Beirut, Lebanon
- Haematological Scientific Center of Ministry of Healthcare of the Russian Federation, Moscow, Russia
- Centre of Excellence in Thrombosis & Hemostasis, King Saud University, Riyadh, Saudi Arabia
- Dept of Haematology, Ege University Children's Hospital, Izmir, Turkey (Türkiye)
- Centre for Haemostasis & Thrombosis, St Thomas' Hospital, London, United Kingdom

RESULTS

PARTICIPANT FLOW:
Groups:
- Octafibrin: Thirty-three patients were screened and 25 patients received at least one administration of Octafibrin for treatment of bleeding or as surgical prophylaxis. Eight patients received Octafibrin for both bleeding and a surgical procedure. One patient was treated for a surgical procedure only.
  Octafibrin was individually dosed to achieve a recommended target plasma fibrinogen level of 100 mg/dL for minor bleeds/surgery or 150 mg/dL for major bleeds/surgery
Period: Overall Study
Arm/Group | Octafibrin
Started | 25
SAFETY Population (25 patients received at least one administration of Octafibrin.) | 25
FAS-Bleeding Population (Patients received Octafibrin for treatment of bleeding.) | 24
Surgical Prophylaxis Population (Patients received Octafibrin for surgical procedures.) | 9
Completed | 18
Not Completed | 7

BASELINE CHARACTERISTICS:
Population: All patients who received at least one Octafibrin administration during the study.
Groups:
- SAFETY Population: All patients who received at least one Octafibrin administration during the study.
Arm/Group | SAFETY Population
Number analyzed (Participants) | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 6
  Between 18 and 65 years | 19
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.04 (12.95)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11
  Male | 14
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 5
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 19
  More than one race | 0
  Unknown or Not Reported | 1

OUTCOME MEASURES:

1. Primary Outcome: Overall Clinical Assessment of the Haemostatic Efficacy of Octafibrin in Treating the First Documented Bleeding Episode of Each Patient.
Description: The first bleeding episode covers the time period from the first Octafibrin infusion until 24 hours (i.e., 1 day) after the last infusion.
  The investigator's overall clinical assessment of haemostatic efficacy for bleeding was based on a 4 point haemostatic efficacy scale. The final efficacy assessment of each patient was adjudicated by the Independent Data Monitoring & Endpoint Adjudication Committee (IDMEAC).
Time Frame: 24 hours after last infusion for each bleeding episode
Measure: Count of Participants; unit: Participants
Groups:
- Investigator Assessment: Efficacy as assessed by the investigator
- IDMEAC Assessment: Efficacy as assessed by the IDMEAC
Arm/Group | Investigator Assessment | IDMEAC Assessment
Number analyzed (Participants) | 24 | 24
Participants
  Excellent | 19 | 23
  Good | 5 | 1
  Moderate | 0 | 0
  None | 0 | 0
  Missing | 0 | 0
  Overall treatment success | 24 | 24

2. Secondary Outcome: Maximum Clot Firmness (MCF) After Fibrinogen Infusion in Each Documented Bleeding Episode (BE), Measured in Frozen Plasma in a Central Laboratory.
Description: MCF (mm) was determined using ROTEM and was used as a surrogate marker for haemostatic efficacy. ROTEM is a method for the continuous measurement of clot formation and clot firmness. It utilises a mechanical detection system which is based on the ability of the blood or plasma clot to form a mechanical coupling over a distance of 1 mm.
Time Frame: Before first infusion and 1 hour after end of first and last infusion of each documented bleeding episode
Measure: Mean (Standard Deviation); unit: mm
Units Other Than Participants: Bleeding Episodes (BEs)
Groups:
- FAS Bleeding: FAS-Bleeding population (change from pre fibrinogen infusion)
Arm/Group | FAS Bleeding
Number analyzed (Participants) | 24
Number analyzed (Bleeding Episodes (BEs)) | 86
mm | 5.79 (2.53)

3. Secondary Outcome: Fibrinogen Plasma Level
Description: Fibrinogen plasma level was assessed using the Clauss fibrinogen assay
Time Frame: Before (pre-infusion), 1 hour and 3 hours after the end of each subsequent infusion as well as at the time of the overall clinical assessment of haemostatic efficacy (i.e., 24 hours after the last infusion of each documented bleeding episode)
Measure: Mean (Standard Deviation); unit: mg/dL
Units Other Than Participants: BEs
Groups:
- Pre-infusion: FAS-Bleeding population pre-infusion.
- Day 1 Post-infusion 1 h: FAS-Bleeding population, day 1 post-infusion 1h
- Day 1 Post-infusion 3 h: FAS-Bleeding population, day 1 post-infusion 3h
- 1 Day After Last Infusion: FAS-Bleeding population 1 day after last infusion
Arm/Group | Pre-infusion | Day 1 Post-infusion 1 h | Day 1 Post-infusion 3 h | 1 Day After Last Infusion
Number analyzed (Participants) | 24 | 24 | 24 | 24
Number analyzed (BEs) | 88 | 89 | 82 | 84
mg/dL | 0.13 (1.17) | 109.01 (24.38) | 104.46 (21.51) | 70.77 (20.59)

4. Secondary Outcome: Response as Indicated by Incremental in Vivo Recovery (IVR)
Description: Incremental IVR (response): calculated as the maximum increase in plasma fibrinogen (i.e., Clauss data) between pre-infusion and 1 and 3 hours post-infusion, divided by the exact dose of Octafibrin.
Time Frame: Pre-infusion and 1 and 3 hours post-infusion
Measure: Mean (Standard Deviation); unit: mg/dL/(mg/kg)
Units Other Than Participants: BEs
Groups:
- FAS-Bleeding: FAS-Bleeding population
Arm/Group | FAS-Bleeding
Number analyzed (Participants) | 24
Number analyzed (BEs) | 88
mg/dL/(mg/kg) | 1.82 (0.42)

5. Secondary Outcome: Efficacy of Octafibrin for All Bleeding Episodes Collected in the Study
Description: The investigator's overall clinical assessment of haemostatic efficacy for bleeding will be based on a 4-point haemostatic efficacy scale. The final efficacy assessment of each patient will be adjudicated by the Independent Data Monitoring & Endpoint Adjudication Committee (IDMEAC)
Time Frame: 24 hours after last infusion for each bleeding episode
Measure: Count of Units; unit: BEs
Units Other Than Participants: BEs
Groups:
- Investigator: FAS-Bleeding population (all bleeding episodes) as assessed by the investigator
- IDMEAC: FAS-Bleeding population (all bleeding episodes) as assessed by the IDMEAC
Arm/Group | Investigator | IDMEAC
Number analyzed (Participants) | 24 | 24
Number analyzed (BEs) | 89 | 89
BEs
  Excellent | 70 | 81
  Good | 16 | 7
  Moderate | 1 | 1
  None | 0 | 0
  Missing | 2 | 0
  Overall treatment success | 86 | 88

6. Secondary Outcome: Efficacy of Octafibrin in Preventing Bleeding During and After Surgery
Description: The efficacy of Octafibrin will be assessed at the end of surgery by the surgeon and post-operatively by the haematologist using two 4-point haemostatic efficacy scales. An overall efficacy assessment taking both the intra- and post-operative assessment into account will be adjudicated by the IDMEAC
Time Frame: First dose of Octafibrin administered prior to elective surgery to at least 3 post-operative days for minor and 7 post-operative days for major surgeries or last post-operative infusion, whichever comes last
Measure: Count of Units; unit: Surgeries
Units Other Than Participants: Surgeries
Groups:
- Surgeon (Intra-op): Octafibrin efficacy assessed by the surgeon during the operation.
- IDMEAC (Intra-op): Octafibrin efficacy assessed by IDMEAC during the operation.
- Haematologist (Post-op): Octafibrin efficacy assessed by the Haematologist after the operation.
- IDMEAC (Post-op): Octafibrin efficacy assessed by IDMEAC after the operation.
Arm/Group | Surgeon (Intra-op) | IDMEAC (Intra-op) | Haematologist (Post-op) | IDMEAC (Post-op)
Number analyzed (Participants) | 9 | 9 | 9 | 9
Number analyzed (Surgeries) | 12 | 12 | 12 | 12
Surgeries
  Excellent | 11 | 11 | 12 | 11
  Good | 1 | 1 | 0 | 1
  Moderate | 0 | 0 | 0 | 0
  None | 0 | 0 | 0 | 0
  Missing | 0 | 0 | 0 | 0
  Overall treatment success | 12 | 12 | 12 | 12

7. Other Pre Specified Outcome: Analysis of Safety: Immunogenicity Testing for Anti-fibrinogen Antibodies
Description: Immunogenicity testing for the presence of anti-fibrinogen antibodies at Day 14 and Day 30 after the administration of Octafibrin for bleeding. An experimental non-standard ELISA was developed for this study for evaluating anti-fibrinogen antibodies. No specific test was performed to discern for neutralizing antibodies. The clinical implications of the assay results are not known.
Time Frame: Up to 30 days (start of the first Octafibrin infusion until the end of each 30-day observation and follow-up period for on-demand treatment or until the Last Post-Operative Day in surgeries)
Measure: Count of Participants; unit: Participants
Groups:
- Pre-infusion: FAS-Bleeding population, immunogenicity testing prior to infusion.
- Observational Period: FAS-Bleeding population, immunogenicity testing during the observational period.*
Arm/Group | Pre-infusion | Observational Period
Number analyzed (Participants) | 24 | 24
Participants
  Participants with Anti-fibrinogen Antibodies | 4 | 6
  Participants without Anti-fibrinogen Antibodies | 20 | 18

ADVERSE EVENTS:
Time Frame: Up to 30 days (start of the first Octafibrin infusion until the end of each 30-day observation and follow-up period for on-demand treatment or until the Last Post-Operative Day in surgeries).
Description: AEs occurring between the start of the first Octafibrin infusion and the end of each 30-day observation and follow-up period and during the surgical follow-up were recorded as treatment-emergent adverse events (TEAEs). Non-TEAEs were all AEs not falling into the follow-up periods
Groups:
- Safety Population: All patients who received at least one administration of Octafibrin during the study
Arm/Group | Safety Population
All-Cause Mortality (participants affected / at risk) | 0/25
Serious Adverse Events (participants affected / at risk) | 5/25
Other Adverse Events (participants affected / at risk) | 19/25
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=25)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 1 (1)
Ligament sprain (Injury, poisoning and procedural complications) | 1 (1)
Patella fracture (Injury, poisoning and procedural complications) | 1 (1)
Transfusion reaction (Injury, poisoning and procedural complications) | 1 (1)
Accelerated hypertension (Vascular disorders) | 1 (1)
Thrombosis (Vascular disorders) | 1 (1)
Peripheral ischaemia (Vascular disorders) | 1 (1)
Dengue fever (Infections and infestations) | 1 (1)
Hepatitis C (Infections and infestations) | 1 (1)
Haemorrhage intracranial (Nervous system disorders) | 1 (1)
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 (2)
Hypocalcaemia (Metabolism and nutrition disorders) | 1 (1)
Abortion spontaneous (Pregnancy, puerperium and perinatal conditions) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Safety Population (N=25)
Gingival bleeding (Gastrointestinal disorders) | 2 (8)
Vomiting (Gastrointestinal disorders) | 2 (4) — Of these, 3 AEs in 2 patients were deemed to be TEAEs.
Abdominal pain upper (Gastrointestinal disorders) | 1 (1) — This/these were deemed to be a TEAE.
Constipation (Gastrointestinal disorders) | 1 (1) — This/these were deemed to be a TEAE.
Gastritis (Gastrointestinal disorders) | 1 (1)
Lip haemorrhage (Gastrointestinal disorders) | 1 (1)
Rectal haemorrhage (Gastrointestinal disorders) | 1 (1) — This/these were deemed to be a TEAE.
Toothache (Gastrointestinal disorders) | 1 (1)
Limb injury (Injury, poisoning and procedural complications) | 3 (3) — This/these were deemed to be a TEAE.
Procedural pain (Injury, poisoning and procedural complications) | 1 (2) — This/these were deemed to be a TEAE.
Arthropod sting (Injury, poisoning and procedural complications) | 1 (1) — This/these were deemed to be a TEAE.
Contusion (Injury, poisoning and procedural complications) | 1 (1) — This/these were deemed to be a TEAE.
Epicondylitis (Injury, poisoning and procedural complications) | 1 (1) — This/these were deemed to be a TEAE.
Incision site pain (Injury, poisoning and procedural complications) | 1 (1) — This/these were deemed to be a TEAE.
Skin wound (Injury, poisoning and procedural complications) | 1 (1) — This/these were deemed to be a TEAE.
Traumatic haemorrhage (Injury, poisoning and procedural complications) | 1 (1) — This/these were deemed to be a TEAE.
Haemorrhage (Vascular disorders) | 1 (7) — Of these, 1 AE was deemed to be a TEAE.
Hypertension (Vascular disorders) | 2 (2) — Of these, 1 AE was deemed to be a TEAE.
Haematoma (Vascular disorders) | 1 (1) — This/these were deemed to be a TEAE.
Brucellosis (Infections and infestations) | 1 (1)
Pharyngitis (Infections and infestations) | 1 (1) — This/these were deemed to be a TEAE.
Purulent discharge (Infections and infestations) | 1 (1) — This/these were deemed to be a TEAE.
Rash pustular (Infections and infestations) | 1 (1)
Rhinitis (Infections and infestations) | 1 (1)
Tonsillitis (Infections and infestations) | 1 (1) — This/these were deemed to be a TEAE.
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 (4)
Arthralgia (Musculoskeletal and connective tissue disorders) | 2 (2) — Of these, 1 AE was deemed to be a TEAE.
Groin pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Muscle haemorrhage (Musculoskeletal and connective tissue disorders) | 1 (1) — This/these were deemed to be a TEAE.
Ecchymosis (Skin and subcutaneous tissue disorders) | 2 (4)
Drug eruption (Skin and subcutaneous tissue disorders) | 1 (1) — This/these were deemed to be a TEAE.
Skin fissures (Skin and subcutaneous tissue disorders) | 1 (1) — This/these were deemed to be a TEAE.
Skin haemorrhage (Skin and subcutaneous tissue disorders) | 1 (1)
Skin lesion (Skin and subcutaneous tissue disorders) | 1 (1)
Headache (Nervous system disorders) | 1 (1)
Hypoaesthesia (Nervous system disorders) | 1 (1)
Genital lesion (Reproductive system and breast disorders) | 1 (1)
Menorrhagia (Reproductive system and breast disorders) | 1 (1)
Pelvic congestion (Reproductive system and breast disorders) | 1 (1)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 1 (1) — This/these were deemed to be a TEAE.
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Upper respiratory tract infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) — This/these were deemed to be a TEAE.
Asthenia (General disorders) | 1 (1) — This/these were deemed to be a TEAE.
Pain (General disorders) | 1 (1) — This/these were deemed to be a TEAE.
Transaminases increased (Investigations) | 1 (1) — This/these were deemed to be a TEAE.
Depression (Psychiatric disorders) | 1 (1) — This/these were deemed to be a TEAE.
Dysuria (Renal and urinary disorders) | 1 (1) — This/these were deemed to be a TEAE.
Reactive thrombocytosis (Blood and lymphatic system disorders) | 1 (1) — This/these were deemed to be a TEAE.
Phlebitis (Vascular disorders) | 1 (1) — This/these were deemed to be a TEAE.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2014-10-31): https://cdn.clinicaltrials.gov/large-docs/26/NCT02267226/Prot_002.pdf
  • Statistical Analysis Plan (2016-07-11): https://cdn.clinicaltrials.gov/large-docs/26/NCT02267226/SAP_003.pdf